CLINICAL TRIAL: NCT00754351
Title: Docetaxel, Gemcitabine and Bevacizumab as Salvage Therapy for Metastatic Breast Cancer
Brief Title: Docetaxel, Gemcitabine and Bevacizumab for Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, Vassilis Georgoulias, MD, Prof. D. Mavroudis, University Hospital of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.01
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: docetaxel; gemcitabine; bevacizumab; chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Bevacizumab->Docetaxel->Gemcitabine
  Interventions: Drug: Bevacizumab; Drug: Docetaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab (IV) 10 mgr/Kgr on days 1 and 15 every 4 weeks for 6 cycles followed by Bevacizumab (IV) 15 mgr/Kgr on day 1 every 3 weeks until disease progression
  Other Names: Avastin
Drug: Docetaxel — Docetaxel (IV) 65 mg/m2 on days 1 and 15 every 4 weeks for 6 cycles
  Other Names: Taxotere
Drug: Gemcitabine — Gemcitabine (IV) 1500 mg/m2 on days 1 and 15 every 4 weeks for 6 cycles
  Other Names: Gemzar

SUMMARY:
This study will evaluate the efficacy and toxicity of docetaxel, gemcitabine and bevacizumab combination, administered biweekly, as salvage treatment in patients with metastatic and HER2 negative breast cancer.

DETAILED DESCRIPTION:
Docetaxel plus gemcitabine is an active combination in the salvage treatment for metastatic breast cancer. Administered every two weeks, this combination has a favorable toxicity profile, and promising activity in > 1st line treatment for metastatic breast cancer. Recently, initial therapy of metastatic breast cancer with paclitaxel plus bevacizumab demonstrated prolonged progression-free survival, as compared with paclitaxel alone. This study will evaluate the addition of bevacizumab to a biweekly regimen of docetaxel and gemcitabine in the salvage therapy for metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically- confirmed metastatic breast adenocarcinoma
* No HER2 overexpression or gene amplification
* At least one previous chemotherapy regimen for metastatic breast cancer
* Age ≥18 years
* Performance status (WHO) 0-2
* Life expectancy of at least 12 weeks
* Measurable disease as defined by at least 1 bidimensionally measurable lesion ≥ 20 X 10 mm
* Performance status (WHO) 0-2
* Adequate liver function (serum bilirubin <1.5 times the upper normal limit, AST and ALT <2.5 times the upper normal limit in the absence of demonstrable liver metastases, or <5 times the upper normal limit in the presence of liver metastases), adequate renal function (serum creatinine <1.5 times the upper normal limit) and bone marrow ≥ 1,500/mm3, PLT ≥ 100,000/mm3, Hgb ≥ 9 g/dL) function
* Written informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Progressive brain metastases according to clinical or radiological criteria
* Brain metastases without prior radiation therapy
* Radiation therapy within the previous 4 weeks
* Previous radiation therapy to the only measurable lesion
* Proteinuria ≥ 500 mgr of protein daily
* Uncontrolled hypertension
* Documented hemorrhagic diathesis or coagulation disorder
* Cardiovascular disease (class II-IV NYHA congestive heart failure, myocardial infarction within the previous 4 months, unstable angina, LVEF < normal, ventricular arrhythmia, uncontrolled hypertension)
* Thrombotic event within the previous 6 months
* Concurrent use of aspirin > 325 mgr daily, low molecular weight heparin in therapeutic dose, warfarin or acenocoumarol, non-steroid anti-inflammatory agents
* Major surgical procedure within the previous 4 weeks
* Presence of nonhealing wound or fracture
* Peripheral neuropathy > grade 2 according to the NCI CTCAE (version 3.0)
* Any sustained chronic toxicity > grade 2 according to the NCI CTCAE (version 3.0)
* Uncontrolled infection
* Any serious, uncontrolled comorbidity on the investigator's judgment
* Other cancer within the previous 5 years, except non-melanoma skin cancer and in situ cervical cancer
* Serious psychiatric illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate | up to 6 months

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
Toxicity profile | 21 days
Overall Survival | 1 year
Quality of life assessment | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (2):
- Greece (2):
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli